CLINICAL TRIAL: NCT02034344
Title: Longitudinal Study of Skin And Systemic Biomarkers In Subjects With Active Cutaneous Lupus Erythematosus And In Healthy Volunteers
Brief Title: A Study of Skin and Systemic Biomarkers In Patients With Active Cutaneous Lupus Erythematosus And In Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR102355; NOCOMPOUNDLUP0001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-12-10; First posted 2014-01-13 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Systemic; Lupus Erythematosus, Discoid; Healthy
Keywords: Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Systemic; Lupus Erythematosus, Discoid; Healthy; Active Cutaneous Lupus Erythematosus; Longitudinal Study; Biomarkers; Subacute Cutaneous Lupus Erythematosus; Skin Biopsy
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Systemic; Lupus Erythematosus, Discoid | interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Healthy participants: 20 healthy participants will be enrolled.
  Interventions: Procedure: Skin biopsy; Procedure: Blood collection; Procedure: Urine collection
- Group 2: DLE/SCLE without SLE: 30 participants with Discoid Lupus Erythematosus/Subacute Cutaneous Lupus Erythematosus (DLE/SCLE) without Systemic Lupus Erythematosus (SLE) will be enrolled.
  Interventions: Procedure: Skin biopsy; Procedure: Blood collection; Procedure: Urine collection
- Group 3: DLE/SCLE with SLE: 30 participants with DLE/SCLE with SLE will be enrolled.
  Interventions: Procedure: Skin biopsy; Procedure: Blood collection; Procedure: Urine collection

INTERVENTIONS:
Procedure: Skin biopsy — Participants with LE will have 2 adjacent 4 mm punch biopsies collected from involved and uninvolved skin at one timepoint and again from the involved skin site approximately 12 weeks later. Healthy participants will have 2 adjacent 4 mm punch biopsies taken at one timepoint.
Procedure: Blood collection — Blood for serum analyses will be taken from all participants. Blood for DNA analysis will only be taken from participants who consent to this separately.
Procedure: Urine collection — Urine will be collected from all participants.

SUMMARY:
The purpose of this study is to obtain skin, blood, and urine samples from patients with active cutaneous lupus lesions and from healthy participants.

DETAILED DESCRIPTION:
This is a Phase 0 multi-center and longitudinal study of biomarkers and clinical parameters in patients with lupus erythematosus (LE). Approximately 80 participants (20 healthy participants and 60 patients with LE) will be enrolled. This will include 30 with Discoid Lupus Erythematosus/Subacute Cutaneous Lupus Erythematosus (DLE/SCLE) without Systemic Lupus Erythematosus (SLE), and 30 with DLE/SCLE with SLE. All patients with LE will continue to be managed by their personal physicians per their standard-of-care. Study participants will undergo interventional procedures that include collection of urine, blood samples and skin biopsy. There will be a single sample collection timepoint for healthy participants and two sample collection timepoints for LE patients, separated by approximately 12 weeks. A blood sample for genomic analysis will be collected for research purposes from patients who provide consent and where local regulations permit. The data obtained in this study will be used in the evaluation of new therapies for lupus and may help in developing new treatments. Safety evaluations will include assessment of adverse events, clinical laboratory tests, vital signs, and physical examinations. The total duration of study participation will be approximately 11 days for healthy participants and 95 days for patients with LE.

ELIGIBILITY:
Inclusion Criteria:

* Have Discoid Lupus Erythematosus (DLE) or Subacute Cutaneous Lupus Erythematosus (SCLE) with or without a diagnosis of Systemic Lupus Erythematosus (SLE)
* Active DLE or active SCLE confirmed by histological analysis (for participants with DLE or SCLE without SLE)
* Confirmed diagnosis of SLE using American College of Rheumatology criteria and has current or historical positive antinuclear antibodies (ANA) or anti double-stranded deoxyribonucleic acid (anti-dsDNA) (for participants with DLE or SCLE with SLE)
* An active skin lesion that can be biopsied (for participants with lupus erythematosus)

Exclusion Criteria:

* Known or thought to have a diagnosis of drug-induced lupus
* An active skin disease that is not a manifestation of lupus erythematosus
* Has an acute cutaneous lupus erythematosus rash only
* If taking anti-malarial therapy has not been on a stable dose for at least 8 weeks before Day 1
* Participants treated with greater than 10mg/day of prednisone therapy or equivalent in the last 4 weeks prior to Day 1
* Positive serology for human immunodeficiency virus antibody, hepatitis B virus, or hepatitis C virus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants and participants with Discoid Lupus Erythematosus (DLE)/Subacute Cutaneous Lupus Erythematosus (SCLE) without Systemic Lupus Erythematosus (SLE) and DLE/SCLE with SLE will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The concentration of individual serum biomarkers | Day 1 (for healthy participants); Day 1 and Day 84 (for participants with lupus erythematosus)
  Investigation of pathways which may be dysregulated in cutaneous lupus lesions

SECONDARY OUTCOMES:
The concentration of individual urine biomarkers | Day 1 (for healthy participants); Day 1 and Day 84 (for participants with lupus erythematosus)
  The presence of potential biomarkers of disease activity will be explored in urine.
The concentration of individual skin biomarkers | Day 1 (for healthy participants); Day 1 and Day 84 (for participants with lupus erythematosus)
  The presence of potential biomarkers of disease activity will be explored in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (21):
- United States (9):
  - La Jolla, California
  - Chicago, Illinois
  - Boston, Massachusetts
  - Lansing, Michigan
  - Neptune City, New Jersey
  - Charlotte, North Carolina
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Salt Lake City, Utah
- Germany (2):
  - Berlin
  - Kiel
- Mexico (3):
  - Chihuahua City
  - Jalisco
  - Mexico City
- Poland (3):
  - Gdansk
  - Krakow
  - Wroclaw
- Taiwan (2):
  - Taichung
  - Taipei
- United Kingdom (2):
  - Leeds
  - London